CLINICAL TRIAL: NCT01826162
Title: The Effects of Differential Short Chain Fatty Acid Availability on Human Substrate and Energy Metabolism
Brief Title: Short Chain Fatty Acid Metabolism and Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MEC 11-3-079
Record Dates: First submitted 2013-02-18; First posted 2013-04-08 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Acetates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sigmoidoscopy (Experimental): 2 actetate concentrations and 1 placebo are administered in randomized order after clipping a catheter in the proximal colon (sigmoidoscopy)
  Interventions: Other: acetate or placebo infusion
- colonoscopy (Experimental): 2 actetate concentrations and 1 placebo are administered in randomized order after clipping a catheter in the distal colon (colonoscopy)
  Interventions: Other: acetate or placebo infusion

INTERVENTIONS:
Other: acetate or placebo infusion

SUMMARY:
Gut microbiota is being increasingly recognized as an important factor in fat distribution, insulin sensitivity and glucose and lipid metabolism. Accordingly, the intestinal microbiota could play an important role in the development of obesity and type 2 diabetes mellitus. The role of gut-derived short-chain fatty acids (SCFA), the formation of which is enhanced by microbial fermentation of fibre, is still controversial. At the present time, our understanding of the effects of SCFA on human metabolism (in gut or systemically) is still limited. The investigators hypothesize that the differential availability of SCFA impacts human metabolism differently.

In this placebo controlled, double-blind, randomized crossover pilot study the investigators will validate in overweight/obese healthy male volunteers whether rectal administration of SCFA is a good model for studying the acute metabolic effects of SCFA. For this, it will be investigated if site of administration (in distal or proximal colon) of SCFA differentially affects parameters of substrate and energy metabolism and to test the duration of short-term effects of SCFA administration.

ELIGIBILITY:
Inclusion Criteria:

* Overweight, obese men

Exclusion Criteria:

* athletes
* diabetes mellitus

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fat oxidation, energy expenditure | 1 study day for each administration
  Fat oxidation and energy expenditure are measured during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load

SECONDARY OUTCOMES:
Hormones that influence substrate and energy metabolism | 1 study day for each administration
  Insulin, Glucagon, GLP-1, PYY and Leptin are measured during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load
Inflammatory markers | 1 study day for each administration
  LBP, TNF-α, IL-6, IL-1 are measured during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load
Plasma SCFA content | 1 study day for each administration
  Plasma SCFA content (acetate, butyrate and propionate) are measured during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load
Circulating metabolites | 1 study day for each administration
  Glucose, FFA, TG, Glycerol, FIAF are measured during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load
Appetite VAS scoring | 1 study day for each administration
  Visual Analogue Scale for hunger and appetite are filled in during fasting acetate/placebo infusion and during acetate/placebo infusion after an oral glucose load

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Blaak, Prof., Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University, Maastricht, Limburg
  - Maastricht University, Maastricht